CLINICAL TRIAL: NCT05396911
Title: Testing an Anti-Tobacco Intervention to Reduce Tobacco and Nicotine Use Among High School Students
Brief Title: Development of UP2UTobacco for High School Youth
Acronym: UP2UTobacco
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Foundation for Healthy Youth (Other)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, Department of Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBS4719
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Cessation; Tobacco Use; Electronic Cigarette Use
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP2UTobacco (Experimental): Youth Brief Tobacco Intervention
  Interventions: Behavioral: UP2UTobacco
- No Treatment Control (No Intervention)

INTERVENTIONS:
Behavioral: UP2UTobacco — The universal prevention program was designed as a group intervention to include components of effective tobacco control programs for youth and young adults. The intervention lasts approximately 45 minutes and is delivered in a classroom setting, utilizing a Socratic teaching style and evoking participation using the principles of motivational interviewing. UP2UTobacco targets all tobacco products with the goals to enhance motivation for youth to quit tobacco or remain tobacco-free, reduce intentions to use tobacco, promote peer discussions around the impact of using tobacco, and correct cognitive misperceptions around tobacco use.
  Other Names: Youth Brief Tobacco Intervention
  Arms: UP2UTobacco

SUMMARY:
Tobacco use is increasing among youth in the U.S. However evidence for the long-term effectiveness of tobacco cessation programs for youth is limited. The current study seeks to adapt and evaluate a universal group-based youth brief tobacco intervention for 9th grade students.

This study will use a sequential, multi-method research design beginning with qualitative roundtable discussions with 9th grade students to adapt an existing young adult brief tobacco intervention for youth. Roundtable discussions with students will identify salient intervention themes and strategies for targeting the intervention and developing the text messages. The second phase of the study evaluates the brief intervention, UP2UTobacco, through a cluster randomized controlled trial that compares UP2UTobacco to a no treatment control. It is hypothesized that the UP2UTobacco will produce greater abstinence at the 6-month follow-up compared to the no treatment control.

Roughly 90% of daily smokers started before the age of 18, and 2,000 youth smoke a cigarette for the first time each day in the U.S. Additionally, e-cigarette use is on the rise among youth, and is linked to cigarette initiation among tobacco naïve youth. In order to curb the rise of tobacco use among youth, interventions that are easily implemented and easily disseminated need to be developed for youth addressing currently available products and contemporary patterns of use. If the interventions in the current study are proven efficacious, they can easily be disseminated to other schools to continue reducing youth tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the selected physical education or health class selected for participation in the study.

Exclusion Criteria:

* None

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 432 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Past 30-day point prevalence abstinence | past 30-day
  The primary outcome measure in this study is self-reported past 30-day abstinence from cigarettes, e-cigarettes, smokeless tobacco, hookah, cigars, little cigars, cigarillos, and pipe tobacco. Past 30-day abstinence will be determined for each product by a "No" response to the question, "In the past 30 days, have you used a <insert tobacco product name>, even one or two times or puffs?"

SECONDARY OUTCOMES:
Past 7-day point prevalence abstinence | past 7 days
  The primary outcome measure in this study is self-reported past 7-day abstinence from cigarettes, e-cigarettes, smokeless tobacco, hookah, cigars, little cigars, cigarillos, and pipe tobacco. Past 7-day abstinence will be determined for each product by a "No" response to the question, "In the past 7days, have you used a <insert tobacco product name>, even one or two times or puffs?"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Little MA, Mallawaarachchi I, Pilehvari A, Velmurugan P, Wester AG, Wiseman KP. Do perceptions of harm and addictiveness influence adolescent's willingness to use various tobacco and nicotine products? Tob Prev Cessat. 2025 Jun 27;11. doi: 10.18332/tpc/204746. eCollection 2025. PMID 40584776